CLINICAL TRIAL: NCT06971146
Title: Health Literacy-Based, Nurse-Led Telehealth Support for Gout Self-Management: the Danish Randomized GOUTCONNECT Trial
Brief Title: Nurse-Led Telehealth for Gout
Acronym: GoutConnect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Silkeborg (Other); Gødstrup Hospital (Other); Randers Regional Hospital (Other); Regionshospitalet Horsens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1-10-72-165-24; 2096-00035B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Health Literacy; Gout Arthritis; Gout Initiating Urate-loweringUrate-lowering Therapy; Telehealth; Digital Health; Adherence
Keywords: self-managment
MeSH Terms: conditions — Arthritis, Gouty

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized controlled superiority trial with two parallel groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led self-management support (Experimental)
  Interventions: Other: Nurse-Led Self-Management Support
- GP-follow up (Active Comparator)
  Interventions: Other: GP-follow up

INTERVENTIONS:
Other: Nurse-Led Self-Management Support — The intervention offers four distinct support options. Patients are free to choose the option that best suits their preferences and needs.
  I1: App-Based Monitoring - Patients receive an app that provides relevant health information, including short educational videos, images, and other resources. Every three months, the app sends a pop-up reminder.
  I2: Reminder by Letter - Patients receive a friendly reminder every three months via e-Boks or postal mail (for those without e-Boks access) encouraging continued treatment adherence.
  I3: SMS Reminder - Patients receive a text message every three months to remind them to continue their treatment.
  I4: Phone Call Check-In - A nurse contacts the patient by phone three times per year at scheduled intervals to provide support and ensure they remain on track with their treatment.
  Arms: Nurse-led self-management support
Other: GP-follow up — Patients in the control group will be discharged from the hospital and continue with routine care provided by their general practitioner (GP). The GP will receive a discharge letter outlining the recommended treatment plan. In addition, patients will receive a letter containing key information about their condition, along with a recommendation to consult their GP annually for ongoing disease monitoring.
  Arms: GP-follow up

SUMMARY:
The aim of this clinical trial is to evaluate whether nurse-led telehealth support helps individuals with gout better manage their condition and adhere to urate-lowering medication after discharge from a rheumatology clinic.

Eligible patients will be recruited from five rheumatology departments in the Central Denmark Region after achieving two consecutive target serum urate levels-below 0.36 mmol/L, or below 0.30 mmol/L for patients with tophi.

Participants will be adults with gout who meet specific medical criteria, are taking medications such as allopurinol or Adenuric, and are able to read and write Danish.

Participants will be randomly assigned to one of two groups:

* Intervention group: nurse-led telehealth support.
* Control group: usual care with follow-up by their general practitioner.

The primary goal is to support patients in maintaining healthy uric acid levels after 52 weeks.

Participants in the nurse-led group have the option to choose from four support options:

I1: App-Based Support - an app provides information and reminders. I2: Letter Reminders - messages are sent via digital or postal mail. I3: Text Reminders - SMS messages are sent every three months. I4: Phone Support - nurses call three times a year to check in.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Fulfills ACR/EULAR 2015 Gout Classification Criteria
* Estimated Glomerular Filtration Rate (e-GFR) >30 ml/min
* Prescribed Allopurinol or Adenuric, and achieved two consecutive serum urate levels of two consecutive serum urate levels of ≤0.30 mmol/l for patients with tophi and ≤0.36 mmol/L for patients without tophi
* Have sufficient Danish reading and writing skills to understand information and complete questionnaires.

Exclusion Criteria:

• Cognitively impaired, unable to understand or provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving target serum urate (s-urate) concentration | 52 weeks
  The number and proportion of participants with a serum urate concentration equal to or less than 0.36 mmol/L or 0.30 mmol/L if tophi, at 52 weeks after randomization.
Gout impact | 52 weeks
  Changes in Gout Impact Scale (GIS). GIS is a patient-reported outcome measure assessing the impact of gout on health-related quality of life. The GIS includes domains such as gout concern overall, gout medication side effects, unmet treatment need, well-being during gout attack, and concern during gout attack. Each domain is scored on a 0-100 scale, with higher scores indicating greater impact (worse health status).
  Change from baseline to week 52 will be calculated, with negative change scores indicating improvement (i.e., reduced gout impact).

SECONDARY OUTCOMES:
Quality of life one year after discharge from a rheumatology clinic indicated by EQ-5D-5L. | 52 weeks
  The EQ-5D-5L is a standardized measure of health status developed by the EuroQol Group, covering five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five levels of severity. An index score will be calculated based on country-specific value sets, with scores typically ranging from <0 (worse than death) to 1 (perfect health). Change from baseline to week 52 will be assessed, with positive changes indicating improvement in health-related quality of life.
Proportion of participants adherent to urate lowering drugs based on CQR-5 | 52 weeks
  Adherence to urate lowering drugs will be assessed using the Compliance Questionnaire Rheumatology 5-item version (CQR-5). The CQR-5 is a patient-reported questionnaire specifically developed to measure adherence in patients with rheumatic diseases. Each item is scored on a 4-point Likert scale, and an overall adherence score is calculated. Participants will be classified as adherent if their CQR-5 score is above the predefined threshold for good adherence (e.g., ≥80% predicted probability of adherence based on validated cutoff.)

OTHER OUTCOMES:
Need for acute healthcare visits | 52 weeks
  The difference in need for acute visits at rheumatologists of rheumatology nurses at the rheumatology department.
All contacts to the rheumatology department | 52 weeks
  The total number of contacts (in-person visits, telephone consultations, video consultations, and written communications) between participants and the rheumatology department during the 52 weeks follow-up period. Contacts include both scheduled and unscheduled interactions related to the management of gout.
Change in Gout-related Global Assessment (PGA) score | 52 weeks
  The Patient Global Assessment (VAS PGA) will be used to assess the patient's overall assessment of their disease status. The VAS PGA is a self-reported measure, where the participant marks their perceived disease activity on a 100 mm horizontal line, with 0 mm indicating "no disease activity" and 100 mm indicating "worst possible disease activity." Change from baseline to 12 months will be assessed, with a lower score indicating a reduction in perceived disease severity.
Change in Health Assessment Questionnaire Disability Index (HAQ-DI) score | 52 weeks
  The Health Assessment Questionnaire Disability Index (HAQ-DI) will be used to assess functional disability in participants with gout. The HAQ-DI consists of 20 questions across 8 domains, including dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Each question is scored from 0 (no difficulty) to 3 (unable to perform), with a higher score indicating greater disability. Change in HAQ-DI score from baseline to 12 months will be assessed, with a reduction in score indicating improvement in functional status.
Number of gout flares | 40 and 52 weeks
  The total number of gout flares experienced by each participant during the 52 week follow-up period. A gout flare is defined as a self-reported episode of acute joint pain, swelling, and/or erythema consistent with gout.
Change in gout related pain measured by Visual Analog Scale (VAS) | 40 and 52 weeks
  Gout related pain will be assessed using a Visual Analog Scale (VAS), where participants rate their current level of pain on a 100 mm horizontal line ranging from 0 mm ("no pain") to 100 mm ("worst imaginable pain"). Change from baseline to 52 week will be calculated, with negative changes indicating a reduction in pain intensity

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Aarhus University Hospital, Aarhus
  - Gødstrup Hospital, Herning
  - Horsens Hospital, Horsens
  - Randers Hospital, Randers
  - Silkeborg Hospital, Silkeborg

IPD SHARING:
Plan to Share IPD: No